CLINICAL TRIAL: NCT05832229
Title: Liver Cirrhosis Network (LCN) Rosuvastatin Efficacy and Safety for Cirrhosis in the United States (RESCU): A Double-Blind Randomized, Placebo-Controlled Phase 2 Study
Brief Title: Liver Cirrhosis Network Rosuvastatin Efficacy and Safety for Cirrhosis in the United States
Acronym: LCN RESCU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The Cleveland Clinic (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); Duke University (Other); Mayo Clinic (Other); University of Miami (Other); University of Michigan (Other); University of California, San Diego (Other); University of California, San Francisco (Other); LAC+USC Medical Center (Other); Virginia Commonwealth University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Cancer Institute (NCI) (NIH); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00070580; 5U24DK130164-04 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis; Cirrhosis, Liver; Cirrhosis Early; Cirrhosis Due to Hepatitis B; Cirrhosis Advanced; Cirrhosis Infectious; Cirrhosis Alcoholic; Cirrhosis Due to Hepatitis C
Keywords: Cirrhosis; Liver; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Fibrosis; Liver Cirrhosis; Liver Cirrhosis, Alcoholic; Non-alcoholic Fatty Liver Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled Phase 2 clinical trial, of 20mg (or 10mg for participants of East Asian ancestry) of rosuvastatin by mouth, once daily. Participants will be randomized (1:1) to either once daily placebo or once daily rosuvastatin.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drug manufacturer and bottler will be unblinded, as will a few members of the Scientific and Data Coordinating Center. All other study team members will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Open-label lead-in period of 4 weeks on 20 mg (10 mg for participants of East ancestry or on a protease inhibitor) rosuvastatin by mouth once daily, followed by a period of 96 weeks rosuvastatin 20 mg daily (10 mg daily for participants of East-Asian ancestry or on a protease inhibitor).
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Open-label lead-in period of 4 weeks on 20 mg (10 mg for participants of East ancestry or on a protease inhibitor) rosuvastatin by mouth once daily, followed by a period of 96 weeks placebo.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Patients meeting all eligibility criteria will be assigned to a randomization arm prior to initiation of a 4-week lead-in phase of the study. All participants will undergo a 4-week, open-label active run-in phase to evaluate initial safety and adherence to rosuvastatin. During this active run-phase, all participants will receive target dose rosuvastatin-- 20 mg daily (10 mg daily for participants of East-Asian ancestry or on a protease inhibitor). After the active run-in phase, all participants will continue with their pre-assigned randomization (1:1) treatment of rosuvastatin 20 mg daily (10 mg daily for participants of East-Asian ancestry or on a protease inhibitor) or matching placebo.
  Other Names: Rosuvastatin 20 mg; Rosuvastatin 10 mg

SUMMARY:
This is a double-blind, phase 2 study to evaluate safety and efficacy of rosuvastatin in comparison to placebo after 2 years in patients with compensated cirrhosis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled Phase 2 clinical trial, of 20mg (or 10mg for participants of East Asian ancestry) of rosuvastatin by mouth, once daily. Participants will be randomized (1:1) to either once daily placebo or once daily rosuvastatin.

Patients meeting all eligibility criteria will be assigned to a randomization arm prior to initiation of a 4-week lead-in phase of the study. All participants will undergo a 4-week, open-label active run-in phase to evaluate initial safety and adherence to rosuvastatin. During this active run-phase, all participants will receive target dose rosuvastatin-- 20 mg daily (10 mg daily for participants of East-Asian ancestry). After the active run-in phase, all participants will continue with their pre-assigned randomization (1:1) treatment of rosuvastatin 20 mg daily (10 mg daily for participants of East-Asian ancestry) or matching placebo.

The total duration of the study will be 96 weeks in the assigned treatment arm plus the 4-week lead-in period. The primary outcome will be the mean change in liver stiffness from the baseline measurement to the end of study liver stiffness, as measured by ultrasound-based vibration-controlled transient elastography (VCTE).

There are 10 participating clinical centers, and we anticipate a total of 256 patients will be recruited for the initial lead-in as we estimate 20% of participants may dropout after the lead-in (256 x 0.8 = 204 for randomization into the study drug treatment phase).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Cirrhosis due to nonalcoholic steatohepatitis, alcohol-associated liver disease, or chronic viral hepatitis (treated hepatitis B virus or hepatitis C virus)
3. Clinical diagnosis of cirrhosis as defined investigator confirmation and the following:

   1. At least one liver biopsy within 5 years prior to consent showing either: Metavir stage 4 fibrosis; Ishak Stage 5-6 fibrosis, OR
   2. At least 2 of the following:

   i. Evidence on imaging: Nodular liver with either splenomegaly or recanalized umbilical vein within the past 48 weeks ii. Liver stiffness: vibration-controlled transient elastography within 48 weeks prior to consent or during Screening ≥15 kilopascal or magnetic resonance elastography within 48 weeks prior to consent or during Screening ≥5 kilopascal iii. Evidence of varices demonstrated on imaging or endoscopy within 3 years prior to consent or during Screening iv. Either: Fibrosis-4>2.67 or platelets <150/mL within 6 months prior to consent or during Screening
4. Two measures of vibration-controlled transient elastography: one at screening and one at the randomization study visit, meeting the following criteria:

   1. The first measure must be ≥ 15 kilopascal.
   2. The two measures must be at least 2 hours apart and no more than 60 days apart from one another.
   3. The mean of two measurements must be ≥ 15 kilopascal.
   4. Additionally, both screening and open-label dispense liver stiffness measures must be ≤50 kPa
5. Compensated defined by:

   1. Absence of ascites/hydrothorax, hepatic encephalopathy or variceal bleeding currently or in the last 48 weeks, as determined clinically by investigator.
   2. If prior history of decompensation, must be without current symptoms of decompensation and no longer requiring treatment of complications for the last 48 weeks, including the use of diuretics for the treatment of ascites, and/or rifaximin or lactulose for the treatment of hepatic encephalopathy. Use of non-selective beta blockers will be allowed.
   3. Child-Pugh score <8
6. Provision of written informed consent.

Exclusion Criteria:

1. Currently on a statin or any statin exposure within 24 weeks prior to consent.
2. Known indication for statin therapy, defined as:

   1. Prior peripheral vascular, cardiovascular or cerebrovascular event for which statins are indicated for secondary prevention, OR
   2. Documented familial hypercholesterolemia, heterozygous familial hypercholesterolemia, OR
   3. Fasting LDL-C ≥ 190 mg/dL
3. Myocardial infarction, Unstable angina, transient ischemic events, or stroke within 24 weeks of screening.
4. Alcohol Use Disorder Identification Test (AUDIT) total score of ≥8 at screening.
5. Patients with limitations in attending study visits.
6. Prisoners.
7. Known prior or current hepatocellular carcinoma (HCC) or cholangiocarcinoma.
8. Known transjugular intrahepatic portosystemic shunt (TIPS), balloon retrograde transvenous obliteration (BRTO) or porto-systemic shunt surgery regardless of time of occurrence.
9. Current (in past 24 weeks prior to consenting) use of medications known to cause hepatic fibrogenesis or confound endpoint assessment, defined as:

   1. amiodarone
   2. methotrexate
   3. warfarin
10. Current (in past 24 weeks prior to consenting) use of medications which may increase risk for rosuvastatin-related myositis or DILI, defined as:

    1. fenofibrate
    2. erythromycin
    3. gemfibrozil
    4. niacin (500 mg or more)
    5. HIV protease inhibitors (darunivar, indinavir, nelfinavir, amprenavir) in patients of East Asian descent
    6. colchicine
    7. cyclosporin
    8. Additional medications that will be excluded:

    atazanavir/ritonavir capmatinib darolutamide dasabuvir/ombitasvir/paritaprevir/ritonavir ledipasvir/sofosbuvir elbasvir/grazoprevir erythromycin glecaprevir/pibrentasvir lopinavir/ritonavir regorafenib ritonavir, in any combination simeprevir sofbuvir/velpatasvir/voxilaprevir sofosbuvir/velpatasvir tafamidis teriflunomide

    *If exposure was for 7 or less days for one of these medications can consider enrollment after 28 days from final dose.
11. Presence of portal or hepatic vein thrombosis
12. Diagnosis of untreated hypothyroidism or on unstable treatment regimen for hypothyroidism
13. Receiving an elemental diet or parenteral nutrition
14. Chronic pancreatitis or pancreatic insufficiency
15. Etiology of cirrhosis other than ALD, NAFLD, or viral hepatitis (excluded diagnoses include cryptogenic immune-mediated such as AIH, PSC and PBC, cardiac cirrhosis or Fontan-associated liver disease, A1AT, Wilson's disease, etc.)
16. Conditions which may confound study outcome:

    1. Unstable or active inflammatory bowel disease
    2. Active infection
    3. Any malignant disease (other than squamous or basal cell carcinoma of the skin) within previous 3 years
    4. Prior solid organ or hematopoietic cell transplant
    5. Bariatric surgery in the last 24 weeks prior to consent or planned bariatric surgery within the next 96 weeks
    6. Current liver-unrelated end-stage organ failures such as end-stage renal disease on dialysis, stage 3-4 congestive heart failure (CHF), current chronic obstructive pulmonary disease (COPD) on home oxygen.
17. Known current medical or psychiatric conditions which, in the opinion of the investigator, would make the participant unsuitable for the study for safety reasons or interfere with or prevent adherence to the protocol.
18. The following laboratory abnormalities within 90 days of screening:

    1. Hemoglobin <10 g/dL
    2. Albumin <3.0 g/dL
    3. Prolonged international normalized ratio (INR) >1.5
    4. Total bilirubin ≥ 2.0 mg/dl (unless due to Gilbert's syndrome or hemolysis as denoted by normal direct bilirubin fraction)
    5. Direct bilirubin ≥ 0.9
    6. Uncontrolled diabetes (HbA1c ≥ 9.5%) within past 90 days.
19. Kidney function abnormalities including:

    1. Dialysis
    2. Baseline eGFR < 30 cc/min with CKD-Epi equation
    3. Known nephrotic proteinuria, defined as 3g or greater of protein in 24-hour urine collection
20. Recent (within 48 weeks) or present hepatic decompensation with ascites/hydrothorax, hepatic encephalopathy or variceal bleeding
21. Untreated chronic hepatitis B or C infection

    1. HCV eligible for enrollment if HCV RNA negative at baseline or documentation of prior SVR12
    2. HBV eligible if an HBV DNA <100 IU/mL within the last 48 weeks and on treatment
22. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 200 U/L, or alkaline phosphatase (ALP) ≥ 300 within the past 24 weeks.
23. Documented history of intolerance to statins
24. Serious comorbid medical disease which in the investigator's opinion renders a life-expectancy less than 96 weeks
25. Active illicit substance use (other than THC), including inhaled or injected drugs, in the 24 weeks prior to screening
26. Pregnancy, planned pregnancy or breastfeeding
27. Current participation in active medication treatment trials (within 24 weeks prior to randomization) or planned participation in active medication treatment trials simultaneous to participation in present trial.
28. Significant existing muscle pain or tenderness or prior history of myasthenia gravis as determined by a site physician.
29. Failure or inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in liver stiffness | 96 weeks
  Mean change in liver stiffness as measured in kilopascal with Vibration-Controlled Transient Elastography between study entry and week 96. Range: 2 to 75 kilopascal. Higher stiffness indicates increased disease progression

SECONDARY OUTCOMES:
Time to disease progression | 96 weeks
  Time to disease progression defined as time to development of decompensation event (ascites, hepatic encephalopathy, variceal bleed) or hepatocellular carcinoma. Analyzed as time-to-event; binary if low counts.
All-cause mortality | 96 weeks
  All-cause mortality: time-to-event, binary if low counts
Time to development of ascites | 96 weeks
  Ascites: time-to-event, binary if low counts
Time to development of overt hepatic encephalopathy | 96 weeks
  Time to development of overt hepatic encephalopathy: time-to-event, binary if low counts
Time to development of variceal bleed | 96 weeks
  Variceal bleed: time-to-event, binary if low counts
Time to development of hepatocellular carcinoma | 96 weeks
  Hepatocellular carcinoma: time-to-event, binary if low counts
Change in spleen stiffness as measured by Vibration-Controlled Transient Elastography (VCTE) | 96 weeks
  Units: kilopascal; Range: 5 to 100 kilopascal; higher stiffness indicates increased disease progression
Change in Child-Turcotte-Pugh score | 96 weeks
  Ordinal score from 5 to 15; higher score indicates further disease progression
Change in Model for End Stage Liver Disease - Sodium (MELD-Na) | 96 weeks
  Unitless; Range: 6-40; higher score indicates further disease progression
Change in liver stiffness via Magnetic Resonance Elastography | 96 weeks
  Units: kilopascal; Range: 0 to 20; higher stiffness indicates increased disease progression
Change in Enhanced Liver Fibrosis test | 96 weeks
  Unitless; Range: 5 to 11; Higher score is worse
Change in Fibrosis-4 | 96 weeks
  Unitless; Range: 0 to 10; higher score indicates more stiffness
Change in patient-reported quality of life scores | 96 weeks
  Patient Reported Outcomes Measurement Information System (29-item version) Global Health T-Score: Population centered at 50 points, standard deviation of 10 (higher score signifies "better" health)
Rate of adverse events | 96 weeks
  Count
Rate of serious adverse events | 96 weeks
  Count
Rate of adverse events of special interest | 96 weeks
  Rate of adverse events of special interest (myopathy, drug-induced liver injury, cardiovascular events, cancer other than hepatocellular carcinoma, new onset diabetes as separate outcomes): Count
Time to cardiovascular events | 96 weeks
  Cardiovascular events: time-to-event, binary if low counts
Time to new onset diabetes | 96 weeks
  New onset diabetes: time-to-event, binary if low counts

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Smith, PhD, Principal Investigator — Northwestern University
Locations (13):
- United States (13):
  - University of California San Diego NAFLD Research Center, La Jolla, California
  - Keck Medical Center of USC, Los Angeles, California
  - LAC + USC Medical Center, Los Angeles, California
  - UCSF/Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - University of Miami Health System, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian/Weill Cornell, New York, New York
  - Columbia University Iriving School of Medicine, New York, New York
  - Duke Liver Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Dataset with National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Repository.
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: Information about the study — http://www.lcnstudy.org